CLINICAL TRIAL: NCT06194422
Title: Psychiatric Comorbidities in Children With Generalized Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Gamal Hashem, resident doctor, Assiut University
Other Study IDs: psychiatric change in children
Record Dates: First submitted 2023-11-20; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Psychiatric Comorbidities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epilepsy is defined as a chronic disorder that presents with recurrent episodes of unprovoked seizures. Epileptic seizures are caused by excessive excitation of cortical neurons. The condition has various etiologies and comorbidities.

Classification;

The Classification of Epilepsies includes several diagnostic levels (steps):

1. from seizure type to epilepsy type (generalized/focal/combined generalized and focal/unknown)
2. etiology (genetic/ structural/ infectious/ metabolic/ immune/unknown). A clinician can use any level of the classification

DETAILED DESCRIPTION:
Epilepsy is defined as a chronic disorder that presents with recurrent episodes of unprovoked seizures. Epileptic seizures are caused by excessive excitation of cortical neurons. The condition has various etiologies and comorbidities Classification

The Classification of Epilepsies includes several diagnostic levels (steps):

1. from seizure type to epilepsy type (generalized/focal/combined generalized and focal/unknown)
2. etiology (genetic/ structural/ infectious/ metabolic/ immune/unknown). A clinician can use any level of the classification. Seizures are classified by the onset (focal, generalized or unknown). All types of seizures can be motor or nonmotor.

Focal seizure may evolve to bilateral tonic-clonic (previously called secondary-generalized). Atonic, clonic, tonic, myoclonic seizures and epileptic spasms can be either of focal or generalized onset.

Unclassified type of seizure was introduced. Most common psychiatric manifestations ; Common psychiatric disorders that have been reported among patients with un controlled generalized epilepsy include :

1. Anxiety.
2. Depression.
3. Attention-deficit hyperactivity disorder.
4. Autism. Psychological distress may be the strongest predictor of health-related quality of life, even including seizure frequency and severity , employment or driving status. Affective disorders are overrepresented in epilepsy, and people with epilepsy may be at risk of dropping out from school. The aim of the present study was to assess factors influencing high school dropout, anxiety, and depression in genetic generalized epilepsy (GGE). Potential predictors of high school dropout were analyzed with logistic regression. Having felt excluded because of epilepsy was significantly associated with high school dropout The issue of stigma in epilepsy must be thoroughly addressed in comprehensive care and may be as important as seizure control when it comes to education and quality of life Attention deficit is one of the most frequent symptoms in children with idiopathic generalized epilepsy (IGE).

However, it is unknown whether this is a global attention deficit or a deficit in a specific attention network. We used the attention network test (ANT) in children with IGE, who were not being treated with antiepileptic drugs (AEDs), to determine the efficiencies of three independent attention networks (alerting, orienting, and executive control). Children with IGE showed a significant deficit in their executive control network and in overall reaction time. However, they did not show any deficit in their alerting or orienting networks. These results suggest that IGE specifically affects the executive control network. Autism spectrum disorders (ASD) are neurodevelopmental disorders typically diagnosed in childhood, characterized by core social dysfunction, rigid and repetitive behaviors, restricted interests, and abnormal sensorial sensitivity. ASD associated with neurological conditions: the co-occurrence of epilepsy is well documented and there is also evidence of a higher prevalence of EEG abnormalities with 4-86% of individuals with ASD presenting epileptiform or not epileptiform EEG abnormalities. The presence of epilepsy in people with ASD may be determined by several structural alterations, genetic conditions, or metabolic dysfunctions, known to play a role in the emergence of both epilepsy and autis

ELIGIBILITY:
Inclusion Criteria:

1. Patients with generalized epilepsy either new or old ,controlled or un controlled .
2. School aged patients (from 6 years to 17 years).
3. Patients on anti epileptic treatment .
4. Patients attending children's neurological unit .

Exclusion Criteria:

1. - children with other types of epilepsy .
2. -children with cerebral palsy.
3. -children with neurodegenerative disease.
4. -children with neurometabolic disease.
5. -mentally retarded children.

Ages: 6 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: psychiatric comorbidities in children with generalized epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-24 (Estimated)

PRIMARY OUTCOMES:
Psychiatric comorbidities in children with generalized epilepsy | baseline
  Measuring the prevalence of ADHD and Autism among children suffering from generalized epilepsy .All cases included in the study will be evaluated by:
  * full history including neurological history .
  * full examination including neurological examination .
  * Investigations:
  * EEG
  * ADHD Symptom Checklist-4 (ADHD-SC4( [8]
  * Gilliam Autism Rating scale ( GARS) [9]
  Sample size calculation:
  Based on determining the main outcome variable, the estimated minimum required total sample size is 62 participants .
  Main outcome variable: to evaluate phsycatric complications among epilitic pediatric patients. based on previous study, (40%) and (11-30%) ADHD and Autisim In epilitic children respectively . [10-11] Main statistical test is chi square to detect the difference in percentage of physiatric disorders( ADHD and Autism) in the two groups . Alpha error = 0.05 Power = 0.80 Allocation ratio= 1 One tailed.